CLINICAL TRIAL: NCT03788109
Title: The Relationship Between Gastric Accommodation, Transient Lower Esophageal Sphincter Relaxations and Reflux Events in Healthy Subjects and in Gastro-esophageal Reflux Disease Patients With or Without Overlapping Dyspepsia
Brief Title: Relationship Between Gastric Accommodation, TLESRs and Reflux in HV and in GERD With or Without Overlapping Dyspepsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S57615
Record Dates: First submitted 2016-07-25; First posted 2018-12-27 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Gastro-esophageal Reflux Disease; Functional Dyspepsia; Health
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- device: combined solid state HRiM (Other): combined solid state high resolution esophageal impedance and manometry (HRiM)
  Interventions: Procedure: device: combined solid state HRiM

INTERVENTIONS:
Procedure: device: combined solid state HRiM — The HRiM catheter (Medical Measurement Systems, Enschede, The Netherlands) incorporating 36 pressure sensors, spaced at 2 cm in the stomach and esophagus and at 1 cm in the LES and upper esophageal sphincter (UES), and 16 impedance channels throughout the esophagus, will be placed transnasally, after topical anesthesia. Manometry will be used to record pressures in the stomach, the esophagus, the LES and the UES. In this way, it is possible to detect and characterize TLESRs, and to measure GA. The impedance channels will be used to measure bolus movement, and thus to detect and characterize gastro-esophageal reflux.

SUMMARY:
Our group recently studied the relationship between intra-gastric pressure (IGP) and reflux events after a meal, both in gastro-esophageal reflux disease (GERD) and in healthy volunteers (HV). Ingestion of a meal was accompanied by a drop in IGP, probably representing gastric accommodation (GA). However, the magnitude of this IGP drop varied, and was inversely correlated with the number of transient lower esophageal sphincter relaxations (TLESRs) and the number of reflux events, both in patients and in HV: a smaller meal-induced drop in IGP was associated with a higher rate of reflux events, and vice versa. These findings suggest that impaired GA is a trigger for reflux. Furthermore, impaired GA is a well-established mechanism underlying symptom generation in functional dyspepsia (FD). Hence, the investigators hypothesize that impaired GA is an important pathophysiological feature explaining the overlap between GERD and FD. To evaluate this hypothesis, the investigators will study the relationship between GA, TLESRs and reflux events in HV and in a group of GERD patients which will be categorized as pure GERD or GERD/FD overlap.

DETAILED DESCRIPTION:
1. INTRODUCTION Gastro-esophageal reflux (GER), the retrograde flow of gastric contents in the esophagus, is a physiologic phenomenon. However, when GER causes symptoms (heartburn/regurgitation) or lesions (esophagitis/Barrett's esophagus), it is referred to as gastro-esophageal reflux disease (GERD). GERD is a highly prevalent condition, occurring in up to 20% of the Western population. Gastric acid has been considered the main pathological factor in GERD and the development of proton pump inhibitors (PPIs), reducing gastric acid secretion, was a major break-through in GERD treatment. However, a large number of GERD patients remain symptomatic in spite of PPI therapy. Combined pH-impedance recordings identified ongoing weakly acidic reflux as the major factor underlying these refractory GERD symptoms. One therapeutic option to eliminate also weakly-acidic reflux is anti-reflux surgery, but this is not devoid of side-effects and has a higher risk of unfavorable outcome in refractory GERD. Hence, intense research was devoted to drugs inhibiting all types of reflux by controlling transient lower esophageal sphincter relaxations (TLESRs), the main mechanism underlying reflux. TLESRs are relaxations of the lower esophageal sphincter (LES) that are not triggered by swallowing and allow reflux of ingested air and gas during belching. They occur mainly postprandially and are triggered by gastric distension, which activates mechanoreceptors in the proximal stomach and a vago-vagal pathway resulting in release of nitric oxide at the LES. Although TLESR frequency is similar in GERD and healthy volunteers (HV), the selectivity of TLESRs to gas reflux is lost in patients and liquid reflux is more likely to occur.

   Pharmacological approaches to inhibit TLESRs, more specifically gamma-aminobutyric acid-B (GABA-B) receptor agonism and metabotropic glutamate receptor type 5 (mGLUR5) antagonism, were evaluated in larger-scale clinical trials. Short-term proof-of-principle studies showed the ability of these agents to increase postprandial LES pressure, inhibit TLESRs and decrease the number of reflux events. Clinical trials mainly evaluated the use of these drugs as add-on therapy in refractory GERD, but all trials failed to show substantial improvement in control of persisting reflux symptoms, with both agents over placebo. Two main problems were identified: 1) these drugs inhibited neurotransmission in the vago-vagal reflex pathways controlling TLESRs. However, it seems that parallel pathways using multiple neurotransmitters exists, as inhibition of TLESRs and reflux events with both agents was in the range of 30-50%; 2) it was suggested that these trials failed to distinguish between ongoing GERD symptoms and functional dyspepsia (FD) symptoms, and that only the former were likely to respond to reflux inhibition.

   FD is one of the most common gastrointestinal (GI) disorders and is defined by the Rome III criteria as the presence of chronic dyspeptic symptoms in the absence of underlying structural or metabolic disease that readily explains the symptoms. Based on these symptoms, the Rome III consensus proposed the subdivision of functional dyspepsia into postprandial distress syndrome (PDS), characterized by postprandial fullness and early satiation, and epigastric pain syndrome (EPS), characterized by epigastric pain or burning. Several studies have established a major overlap between GERD and FD, and against this background overlap of both symptom complexes is not surprising.
2. RATIONALE AND OBJECTIVES Our group recently studied the relationship between intra-gastric pressure (IGP) and reflux events after a meal, both in GERD and in HV. Ingestion of a meal was accompanied by a drop in IGP, probably representing gastric accommodation (GA). However, the magnitude of this IGP drop varied, and was inversely correlated with the number of TLESRs and the number of reflux events, both in patients and in HV: a smaller meal-induced drop in IGP was associated with a higher rate of reflux events, and vice versa. These findings suggest that impaired GA is a trigger for reflux. Furthermore, impaired GA is a well-established mechanism underlying symptom generation in FD. Hence, the investigators hypothesize that impaired GA is an important pathophysiological feature explaining the overlap between GERD and FD. To evaluate this hypothesis, the investigators will study the relationship between GA, TLESRs and reflux events in HV and in a group of GERD patients which will be categorized as pure GERD or GERD/FD overlap.
3. GENERAL DESCRIPTION OF THE STUDY In 20 HV, a combined solid state high resolution esophageal impedance and manometry (HRiM) catheter will be placed into the stomach. The investigators will record 30 min before and 60 min after administration of a high carbohydrate and high fat meal (1000 kcal). Esophageal body contractility, LES pressure, TLESRs and reflux events will be identified and classified using established criteria. The number of TLESRs and the number of reflux events will be counted. In sensors 5 cm below the lower border of LES, the magnitude of the meal-induced drop in IGP (deltaIGP) will be measured. Upper gastrointestinal symptoms will be recorded throughout the studies. These measures will provide normal range reference data for further pathophysiological and mechanistic studies in GERD and FD.

   The same protocol will also be used to study 50 GERD patients who will be categorized as pure GERD or GERD/FD overlap (26). GA, quantified as deltaIGP, and the prevalence of impaired GA will be determined in both groups. The correlation between diagnostic category and size of GA will be evaluated, and the investigators will analyze the presence of a hiatal hernia (HH), esophageal peristalsis, fasting and postprandial LES pressure, occurrence of TLESRs, occurrence and characterization of reflux events and their possible correlation with GA. Based on previous studies in GERD, FD and health, the numbers should be sufficient to detect differences in IGP with a power of 80% at a significance level of 0.05.
4. MATERIALS AND METHODS

STUDY SUBJECTS This study will be performed in 20 HV, and in 25 GERD and 25 GERD/FD overlap patients. All subjects are aged between 18 and 65 years, and will receive and sign a copy of the informed consent, before initiation of the study. Discontinuation of all acid suppressive therapy for at least 7 days is mandatory in all patients.

--> HEALTHY VOLUNTEERS

Exclusion criteria:

* history of any upper gastrointestinal (GI) symptoms or GI surgery;
* psychological disorders;
* any drug history;
* use of medication altering GI motility;
* pregnant or nursing women.

  * GERD PATIENTS

Inclusion criteria:

* typical symptoms of reflux, such as heartburn and/or regurgitation;
* gastro-esophageal reflux assessed by 24-h pH-impedance monitoring or a positive symptom association or;
* esophagitis assessed by upper GI endoscopy with careful evaluation of the presence and extent of a hiatal hernia (HH).

Exclusion criteria:

* psychological disorders;
* any drug history;
* use of medication affecting GI motility;
* pregnant or nursing women;
* history of GI surgery.

  -->DETECTION OF FD OVERLAP IN THE GERD POPULATION
* FD symptoms according to the Rome III criteria. The symptoms of FD include one or more of: bothersome postprandial fullness occurring after normal sized meals, early satiation that prevents finishing a regular meal, epigastric pain, and epigastric burning at least several times per week during the last 6 months.
* The investigators will stratify to have equal numbers of overlap and non-overlap patients.

STUDY PROTOCOL Patients and volunteers will be fasted for at least 12 h before the manometry study. Furthermore, they will be asked to refrain from alcohol, tea and coffee at least 12 h before participation, and to refrain from smoking cigarettes at least 1 h before the start of the experiment.

The HRiM catheter (Medical Measurement Systems, Enschede, The Netherlands) incorporating 36 pressure sensors, spaced at 2 cm in the stomach and esophagus and at 1 cm in the LES and upper esophageal sphincter (UES), and 16 impedance channels throughout the esophagus, will be placed transnasally, after topical anesthesia. Manometry will be used to record pressures in the stomach, the esophagus, the LES and the UES. In this way, it is possible to detect and characterize TLESRs, and to measure GA. The impedance channels will be used to measure bolus movement, and thus to detect and characterize gastro-esophageal reflux.

Patients and volunteers will be studied in a semi-recumbent fashion for a 5-10 min stabilization period after the placement of the catheter. Thereafter, subjects will be given 10 wet swallows of 5 ml saline to study esophageal peristalsis. Recordings will be made for 30 minutes after which all subjects will receive a high carbohydrate and high fat meal of 1000 kcal (mashed potatoes, meatloaf, and apple sauce). After meal ingestion, subjects will be monitored for 5 h, after which the catheter will be removed.

ELIGIBILITY:
Inclusion Criteria:

* GERD patients:

  * typical symptoms of reflux, such as heartburn and/or regurgitation;
  * gastro-esophageal reflux assessed by 24-h pH-impedance monitoring or a positive symptom association or;
  * esophagitis assessed by upper GI endoscopy with careful evaluation of the presence and extent of a hiatal hernia (HH).
* GERD/FD overlap:

  * FD symptoms according to the Rome III criteria. The symptoms of FD include one or more of: bothersome postprandial fullness occurring after normal sized meals, early satiation that prevents finishing a regular meal, epigastric pain, and epigastric burning at least several times per week during the last 6 months.

Exclusion Criteria:

* Healthy volunteers:

  * history of any upper gastrointestinal (GI) symptoms or GI surgery;
  * psychological disorders;
  * any drug history;
  * use of medication altering GI motility;
  * pregnant or nursing women.
* GERD patients:

  * psychological disorders;
  * any drug history;
  * use of medication affecting GI motility;
  * pregnant or nursing women;
  * history of GI surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Change in number transient lower esophageal sphincter relaxations | 6-hour study period
  Change in number TLESRs between preprandial and postprandial period

SECONDARY OUTCOMES:
Change in number of reflux episodes | 6 hour study period
  Change in number of reflux episodes between preprandial and postprandial period
Change in intragastric pressure | 6 hour study period
  Change in intragastric pressure between preprandial and postprandial period

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Prof. Dr., Principal Investigator — KULEUVEN, UZLEUVEN
Locations (1):
- Translational Research Center for Gastrointestinal Disorders (TARGID), KU Leuven Campus Gasthuisberg O&N1, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No